CLINICAL TRIAL: NCT01848366
Title: Biowave Overactive Bladder (OAB) Trial
Brief Title: Utilization of the BIOWAVE Device to Treat Overactive Bladder
Acronym: OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth Peters, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Chairman, Department of Urology, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-034
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Overactive Bladder
Keywords: Frequency; urgency; incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biowave Treatment (Experimental): Twelve weekly treatments
  Interventions: Device: Biowave Treatment

INTERVENTIONS:
Device: Biowave Treatment — Twelve weekly treatments

SUMMARY:
Demonstrate a response to stimulation of the posterior tibial nerve using the Biowave device and a microneedle patch electrode in patients with overactive bladder symptoms. The investigators hypothesize that after at least 6 weekly treatments there will be modest improvements in overactive bladder symptoms trending toward more improvement.

DETAILED DESCRIPTION:
Women 18 years old and over with a score of equal to or greater than 4 on the OAB-q short form for urgency and average daily urinary frequency equal to or greater than 10 times based on a 3-day voiding diary plus other inclusion criteria will be reviewed for possible enrollment in this study. Outcomes measured include Global Response Assessment (GRA) for overall bladder symptoms, a change in the 3-day voiding diary parameters and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age
* A score of > 4 on the OAB-q short form for urgency (question 1)
* Average daily urinary frequency > 10 times based on a 3-day voiding diary
* Self-reported bladder symptoms present > 3 months
* Self-reported failed conservative care (i.e., dietary restriction, fluid restriction, bladder training, behavioral modification, pelvic muscle training, biofeedback, etc.)
* Off all antimuscarinics for at least 2 weeks prior to enrollment
* Capable of giving informed consent
* Ambulatory and able to use a toilet independently, without difficulty
* Capable and willing to follow all study-related procedures

Exclusion Criteria:

* Pregnant as confirmed by urine pregnancy test, or plans to become pregnant during the study period
* Neurogenic bladder
* Botox® use in bladder or pelvic floor muscles in the past year
* Pacemakers or implantable defibrillators
* Primary complaint of stress urinary incontinence
* Current urinary tract infection (UTI)
* Current vaginal infection
* Current use of InterStim®
* Current use of Bion®
* Previously been treated with Percutaneous Tibial Nerve Stimulation (PTNS)
* Use of investigational drug/device therapy within the past 4 weeks.
* Participating or have participated within the past 4 weeks in any clinical investigation involving or impacting gynecologic, urinary or renal function.
* Deemed unsuitable for enrollment in study by the investigators based on subjects' history or physical examination (including skin disorders at the treatment site or peripheral neuropathy).
* Subjects with nerve damage that would impact either percutaneous tibial nerve or pelvic floor function.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biowave Treatment
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biowave Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 56.6 [43 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Global Response Assessment (GRA)
Description: The GRA will be used to assess for changes in urinary condition and symptoms after 12 weekly BIOWAVE treatments. The GRA asks the participant to indicate how their condition or symptoms have changed compared to when they started the study. Eight questions addressed bladder symptoms, urine leakage related to activity, urine leakage associated with urge, urinary frequency, Interstitial Cystitis/Painful Bladder Syndrome (IC/BPS), fecal incontinence, and irritable bowel syndrome. Responses range from 1=Markedly Worse to 7=Markedly Improved.
Time Frame: 3 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Biowave Treatment
Number analyzed (Participants) | 8
units on a scale
  Bladder Symptoms | 5.25 [4 to 7]
  Urine Leakage with Activity | 4 [4 to 4]
  Urge Incontinence | 4.6 [4 to 6]
  Urinary Frequency | 5.1 [4 to 7]
  Urinary Urge | 4.9 [4 to 7]
  IC/BPS | 4.3 [4 to 5]
  Fecal Incontinence | 4 [4 to 4]
  Irritable Bowel Symptoms | 4.25 [4 to 5]

ADVERSE EVENTS:
Time Frame: 13 Weeks
Arm/Group | Biowave Treatment
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Due to the small number of subjects enrolled, the results of this preliminary study are limited and not generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No